CLINICAL TRIAL: NCT04468529
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Effect of Injectable Neucardin on the Cardiac Function of Subjects With Chronic Systolic Heart Failure on Standard Heart Failure Therapy
Brief Title: Evaluate the Effect of Injectable Neucardin on the Cardiac Function of Subjects With Chronic Systolic Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZS-01-308
Record Dates: First submitted 2020-07-06; First posted 2020-07-13 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2022-02

CONDITIONS: Chronic Systolic Heart Failure
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double-blind, standard therapy based, placebo-controlled parallel study.
Who Masked: Participant
Masking Description: It is planned to conduct the study in several domestic clinical research sites at the same time. A total of 140 subjects will be enrolled, including 70 subjects in the investigational drug group and 70 subjects in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational drug group (Experimental): Injectable Neucardin + standard basic therapeutic medication
  Interventions: Drug: Recombinant human Neuregulin for injection
- Placebo group (Placebo Comparator): placebo + standard basic therapeutic medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant human Neuregulin for injection — 10 hours per day i.v. drip for the first 10 days (0.6ug/kg/day)
  Other Names: Neucardin
  Arms: Investigational drug group
Drug: Placebo — 10 hours per day i.v. drip for the first 10 days (0ug/kg/day)
  Arms: Placebo group

SUMMARY:
A multi-center, randomized, double-blind, placebo-controlled phase III clinical trial to evaluate the effect of injectable Neucardin on the heart function in male patients with NT-proBNP ≤ 1700 pg/ml and female patients with NT-proBNP ≤ 4000 pg/ml, NYHA II-III chronic systolic heart failure, and to confirm its efficacy and safety.

DETAILED DESCRIPTION:
This trial is planned to be conducted simultaneously in multiple domestic clinical research site, and a total of 140 subjects will be enrolled, including 70 subjects in the investigational drug group and 70 subjects in the placebo group.

Primary endpoint: LVESVI change from baseline on day 30 Secondary endpoints: LVEF Change from baseline on day 30 and day 90. LVESV, LVEDV, LVEDVI change from baseline on day 30. LVESV, LVESVI, LVEDV, LVEDVI change from baseline on day 90. NT-proBNP change from baseline on day 30 and day 90. NYHA class change from baseline on day 30 and day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, male or female;
2. Confirmed diagnosis of heart failure, in stable condition currently, NYHA class II-III, left ventricular ejection fraction (LVEF)≤40% (measured by echocardiography with modified Simpson's method at Screening 1, and measured by CMR at Screening 2 and baseline);
3. Male NT-proBNP ≤1700 pg/ml or female NT-proBNP≤4000 pg/ml (detected by Roche kit in the central laboratory at screening 1);
4. Receiving standard basic therapeutic medication for heart failure for more than 3 months, at the target dose or maximum tolerated dose for more than 1 month, or no change in dose within the last 1 month;
5. Understand and sign the informed consent form.

Exclusion Criteria:

1. Atrial fibrillation during the screening period;
2. Conditions limiting CMR examination, such as installation of pacemakers, ICDs, CRTs or other similar devices contraindicated for CMR, or have claustrophobia;
3. Hypertrophic cardiomyopathy with outflow tract obstruction, constrictive pericarditis, significant and uncorrected valvular heart disease (severe regurgitation or severe stenosis or valvular disease requiring surgery), congenital heart disease requiring surgery but not yet undergoing surgical treatment, primary pulmonary hypertension or secondary severe pulmonary hypertension (≥ 70 mmHg);
4. Right heart failure due to lung disease;
5. Subjects with chronic heart failure complicated with acute hemodynamic disturbance or acute decompensation within recent 1 month (symptoms and signs indicate chronic heart failure is aggravated, and intravenous drug therapy may be required);
6. Angina pectoris within 3 months;
7. Myocardial infarction within the past 6 months;
8. Cerebrovascular accident, revascularization (PCI or other surgery), cardiac surgery, carotid artery or other large vessel surgery within the past 6 months;
9. Prepare to install pacemaker, ICD, CRT or other similar devices within 6 months;
10. History of heart transplantation, use of ventricular assist device (VAD) or preparation for heart transplantation, VAD;
11. Diagnosis of peripartum or chemotherapy-induced cardiomyopathy within the past 12 months;
12. Serious arrhythmia (sustained ventricular tachycardia or other conditions meet the criteria according to the investigator's judgement );
13. Clinical diagnosis of pericardial effusion, pleural effusion or B ultrasound showed pericardial effusion (greater than 50ml or 3 mm) or pleural effusion (greater than 200ml or 10 mm);
14. Liver or kidney dysfunction, chronic liver disease may have a potential impact on liver function, non-heart failure induced bilirubin or alkaline phosphatase > 2 times the upper limit of normal, aspartate aminotransferase or alanine aminotransferase > 3 times the upper limit of normal, eGFR calculated using the MDRD method < 30 ml/min/1.73m2 ;
15. Systolic blood pressure < 90 mmHg or > 160 mmHg;
16. Blood K + < 3.2 mmol/L or > 5.5 mmol/L;
17. Subjects with an absolute change in LVEF > 5% as detected by CMR between screening 2 and baseline;
18. Women of childbearing age who are planning to become pregnant within 2 years (women of childbearing age are defined as all women with physiological capability to become pregnant), and pregnant or lactating women;
19. Patients whose survival time is expected to be less than 6 months as judged by the investigator;
20. Those who have participated in any drug clinical trial within the previous 3 months;
21. Severe neurological disorders (Alzheimer's disease, progressive parkinsonism);
22. The subjects with tumor history or is suffering from tumor now, or with precancerous lesions confirmed by pathological examination (such as breast ductal carcinoma in situ, or cervical dysplasia), or with malignant mass found by examination (physical examination, X-ray examination or B ultrasound examination or other means);
23. The subjects with proliferative glands or adenomas that are found to have endocrine activity that affects cardiac function or endocrine function detected by examinations (physical examination, X-ray examination, B ultrasound examination or other means), such as pheochromocytoma, thyromegaly, etc. (patients with euthyroid thyroid or normal thyroid function do not need to be excluded);
24. The subject, in the judgment of the Investigator, is unable to complete the study or to comply with the requirements of the study (for administrative or other reasons).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Left Ventricular End-Systolic Volume Index(LVESVI) change from baseline on day 30 | Day 30
  Left Ventricular End-Systolic Volume Index(LVESVI) change from baseline

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction(LVEF) Change from baseline on day 30 and day 90 | Day 30 and Day 90
  Left Ventricular Ejection Fraction(LVEF) Change from baseline
Left Ventricular End-Systolic Volume Index(LVESVI) change from baseline on day 90 | Day 90
  Left Ventricular End-Systolic Volume Index(LVESVI) change from baseline
Left Ventricular End-Systolic Volume(LVESV)change from baseline on day 30 and day 90 | Day 30 and Day 90
  Left Ventricular End-Systolic Volume(LVESV)change from baseline
Left Ventricular End-Diastolic Volume(LVEDV)change from baseline on day 30 and day 90 | Day 30 and Day 90
  Left Ventricular End-Diastolic Volume(LVEDV)change from baseline
Left Ventricular End-Diastolic Volume Index(LVEDVI )change from baseline on day 30 and day 90 | Day 30 and Day 90
  Left Ventricular End-Diastolic Volume Index(LVEDVI )
N-Terminal pro-Brain Natriuretic Peptide(NT-proBNP) change from baseline on day 30 and day 90 | Day 30 and Day 90
  N-Terminal pro-Brain Natriuretic Peptide(NT-proBNP) change from baseline
New York Heart Association(NYHA) class change from baseline on day 30 and day 90 | Day 30 and day 90
  New York Heart Association(NYHA) class change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xinchun Yang, M.D, Principal Investigator — Beijing Chao Yang Hospital
Locations (29):
- China (29):
  - Beijing Chaoyang Hospital of Capital Medical University, Beijing
  - Beijing Friendship Hospital of Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - Fuwai hospital chinese Academy of Medical Sciences, Beijing
  - China-Japan Union Hospital of Jilin University, Changchun
  - The First Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - Chongqing University Three Gorges Hospital, Chongqing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - First Affiliated Hospital,Sun Yat-sen University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Haikou People's Hospital, Haikou
  - Hainan General Hospital, Hainan
  - Hunan Provincial People's Hospital, Hunan
  - Jinan Central Hospital, Jinan
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Province QianFoshan Hospital, Jinan
  - Luoyang Center Hospital, Luoyang
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing
  - Shanghai First People's Hospital, Shanghai
  - Shanghai JiaoTong University Ruijing Hospital, Shanghai
  - Shanghai Putuo District Central Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - First Hospital of Shanxi Medical University, Taiyuan
  - Shanxi Cardiovascular Hospital, Taiyuan
  - People's Hospital of Tianjin, Tianjin
  - The Second Hospital of Tianjin Medical University, Tianjin
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No
Zensun ensures that the key information about the design of this protocol will be published in a publicly available database such as www.clinicaltrials.gov. After the end of the trial, Zensun will assist the study site to objectively summarize the trial results, use appropriate statistical methods to analyze the trial data, objectively evaluate the safety and efficacy of the drug according to the results, and make a complete written summary report of the clinical trial. Study results will be submitted for publication and/or publication in a publicly available database. If other individuals or institutions related to this study want to publish or publish the study results or related data, they need to obtain the consent of the sponsor in advance. If the sponsor needs to include the name of the investigators in any publication or advertisement, the consent of the investigator should be obtained.